CLINICAL TRIAL: NCT04504552
Title: Phase II Trial, Open Label, Single-arm, of Immune Checkpoint Inhibitor In High Risk Oral Premalignant Lesions
Brief Title: Immune Checkpoint Inhibitor In High Risk Oral Premalignant Lesions
Acronym: IMPEDE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Paolo Bossi, Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPEDE
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Oral Premalignant Lesions
MeSH Terms: interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Avelumab (Experimental): Avelumab monotherapy on the Day 1 (± 2 days) of a 2-week treatment cycle for 4 administrations.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Subjects will receive treatment with avelumab monotherapy 800 mg as a 60-minute IV infusion on the Day 1 (± 2 days) of a 2-week treatment cycle for 4 administrations.
  Other Names: Bavencio

SUMMARY:
This trial is designed as a prospective, multi-centre, open-label, single-arm, phase II study.

Oral Premalignant Lesions (OPL) may be considered the equilibrium phase of the immunoediting concept, i.e. a dynamic process between the tumour cells and the immune system including surveillance by the immune system or tumour progression. Thus, an imbalance in immunosuppressive microenvironment is a possible key in malignant transformation. In this regard, the activation of the PD-1/PD-L1 pathway has a central role, witnessed by the expression of PD-L1 by multiple cell types within the microenvironment of OPL (tumour-associated macrophages, fibroblasts, lymphocytes) and by the fact that PD-L1 expression in epithelial and subepithelial cells is associated with malignant transformation. The use of checkpoint inhibitors in this setting seems to be justified by this rationale. Employing intermediate end-point markers during preventive strategies against OPL may allow the conduction of smaller trials, able to give insights for designing larger studies and to better select the population receiving benefit from the treatment. In this regard, the evaluation of phenotypic changes (reduction in size or in grade of dysplasia) may not be enough to assess the potential benefit of an intervention. Modulation of molecular markers may be more precise indicator of oral cancer risk in patients with OPL. Thus, the change in LOH at critical loci may be considered intermediate end-point biomarkers of prevention as well as predictors of cancer risk at baseline. Previous experience with anti-EGFR agents showed the feasibility of such measures in a prevention trial.

DETAILED DESCRIPTION:
OPL represent the most common oral precancerous condition, with a potential of malignant transformation varying from 1% to 47% in different studies. Among molecular markers, the most effective in predicting oral cancer risk is loss of heterozygosity (LOH), which may appear in tissues with different histological grade of dysplasia. Patients carrying OPL with LOH at 3p14 and/or 9p21 plus LOH at another locus have an expected 3-year risk of developing oral cancer of 35%. This chromosomal profile is found in about 28% of OPL. Moreover, when a patient has previously suffered from oral cavity cancer, the 3-year risk of malignant transformation for OPL with such a chromosomal profile reaches 69%. The presence of tumour suppressor genes (TSGs) at these chromosomal loci explains the potential for cancer development in the presence of such alterations.

The clinical management of small OPL is excision by a cold knife or laser. However, treatment is not effective to prevent oral cancer in patients. Lesions recur frequently and transform subsequently, and tumours develop in the same or adjacent anatomical region. For larger OPL the clinical management is limited to lifelong surveillance. To improve clinical management of OPLs, the arsenal of treatments should be expanded.

Therefore, this study is aimed at treating high-risk OPL with a short course of immunotherapy (avelumab)

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Male or female > 18 years of age;
3. ECOG Performance status (PS) 0-1;
4. Clinical and histological evidence of OPL with high risk of malignant transformation as defined by LOH at 3p14 and/or 9p21 plus at least at one additional chromosomal site (4q, 8p,11p,13q, or 17p) or patients with a prior oral cancer history and LOH at 3p14 and/or 9p21 (LOH defined according to EPOC trial). These conditions define "LOH positivity";
5. OPL with a histological definition of dysplasia and a minimum diameter of at least 20 mm;
6. Be willing to provide tissue from newly obtained oral biopsies;
7. Not receiving chronic systemic steroidal therapy or any immunosuppressive therapy within 7 days prior to the first treatment; absence of active autoimmune disease that required systemic treatment in the past 2 years, except the following:

   * Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra-articular injection);
   * Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent;
   * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication);
8. Adequate bone marrow function: neutrophils > 1.5 x 109/L, platelets > 100 x 109/L, haemoglobin > 9 g/dL;
9. Adequate liver function: bilirubin < 2 X upper normal limit (except known medical reason not interfering with liver function, such as Gilbert disease), SGOT, SGPT, AP, GGT < 3 x ULN;
10. Adequate renal function: calculated or analysed creatinine clearance > 60 mL/min;
11. If of childbearing potential, willingness to use effective contraceptive method (Pearl Index < 1; e.g. oral contraceptive (pill), hormone spiral, hormone implant, transdermal patch, a combination of two barrier methods (condom and diaphragm), sterilization, sexual abstinence for the study duration and 2 months post-dosing.

Exclusion Criteria:

1. Previous immunotherapy (anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint receptors);
2. Oral lesions due to lichen planus;
3. Diagnosis of prior immunodeficiency or organ transplant requiring immunosuppressive therapy, or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness;
4. Any test for hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating acute or chronic infection;
5. Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for the administration of inactivated vaccines (for example, inactivated influenza vaccines);
6. Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months;
7. Significant neurologic or psychiatric disorders including dementia or seizures;
8. Active uncontrolled infection (requiring IV antibiotics) or active tuberculosis;
9. Active disseminated intravascular coagulation;
10. Other serious underlying medical conditions which could impair the ability of the patient to participate into the study;
11. Having participated in another clinical trial or having received any investigational agent in the preceding 30 days before study entry;
12. Known allergic/hypersensitivity reaction to any of the components of the treatment;
13. Pregnancy (absence confirmed by serum/urine beta HCG) or breastfeeding;
14. Other active malignancy within 3 years, with the exception of a history of a previous, adequately treated:

    * basal cell carcinoma of the skin
    * pre-invasive carcinoma of the cervix
    * superficial bladder cancer
    * carcinoma in situ of the prostate, cervix or breast,
    * head and neck squamous cell carcinoma, surgically treated (radiotherapy treatment not allowed);
15. Legal incapacity or limited legal capacity;
16. Medical, psychological or socio-geographical condition or situation which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent;
17. Active, known or suspected autoimmune disease. Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to be enrolled;
18. Conditions requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days of study drug administration. Inhaled or topical steroids, steroids as premedication for hypersensitivity reactions and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival or malignant transformation-free survival | Every 2 weeks for the first 6 months, then every month for 1 year, then every 3 months for 30 months
  Recurrence or malignancy-free survival since immunotherapy start, for which the events of interest are the recurrence of OPL with LOH or malignant transformation of OPL
Change in LOH status (positive to negative) of OPL | 6 months
  Change in LOH status (positive to negative) of OPL after 6 months since the start of immunotherapy. This is defined as disappearance of any high-risk LOH (and the nonappearance of any other high-risk LOH) in the site of the OPL at the histological sample after immunotherapy treatment

SECONDARY OUTCOMES:
Safety of immunotherapy in the treatment of OPL | Through study completion, an average of 5 years
  Grade 3-5 adverse events or any treatment interruption due to toxicities (safety)
Grading of OPL | 6 months
  Change of histological grading of OPL
Multi-omic signatures | 6 months and through study completion, an average of 5 years
  Identification of multi-omic signatures associated with response to immunotherapy

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo, Torino
  - ASST Spedali Civili di Brescia, Brescia
  - IRCSS Ospedale Policlinico San Martino, Genova
  - Istituto europeo di oncologia, Milan
  - Istituto nazionale dei tumori Regina Elena, Roma

IPD SHARING:
Plan to Share IPD: Yes
After the end of the trial, the genomic data of OPL will be made publicly available through GEO
Supporting Information: CSR
Time Frame: 12 months after the end of the trial, for at least 1 year
Access Criteria: NS

REFERENCES:
- [Derived] Gurizzan C, Lorini L, Paderno A, Tomasoni M, Zigliani G, Bozzola A, Ardighieri L, Battocchio S, Bignotti E, Ravaggi A, Romani C, De Cecco L, Serafini MS, Miceli R, Bardellini E, Majorana A, Piazza C, Bossi P. Immunotherapy for the prevention of high-risk oral disorders malignant transformation: the IMPEDE trial. BMC Cancer. 2021 May 17;21(1):561. doi: 10.1186/s12885-021-08297-3. PMID 34001010